CLINICAL TRIAL: NCT02541305
Title: EFFICACY OF AN EXERCISE PROPRIOCEPTIVE PROGRAM ON PREDICTORS OF RISK OF FALLS IN INSTITUTIONALIZED ELDERLY
Brief Title: EFFICACY OF AN EXERCISE PROPRIOCEPTIVE PROGRAM IN INSTITUTIONALIZED ELDERLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Socio- Health Center Puente Real ( Health Care for Older © ) of Badajoz (Unknown)
Responsible Party: Principal Investigator, JOSE VICENTE TOLEDO MARHUENDA, PhD, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JVT001
Record Dates: First submitted 2015-07-31; First posted 2015-09-04 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Accidental Falls
Keywords: falls prevention; proprioception; physical condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cotrol (Active Comparator): No propioceptive program.
  Interventions: Other: No propioceptive program
- Experimental (Experimental): Propioceptive program
  Interventions: Other: propioceptive program

INTERVENTIONS:
Other: propioceptive program — The training program has 6 specific proprioceptive exercises, each five minutes long, which will conducted in static and dynamic positions for a period of 30 minutes. Each exercise session will include 55 minutes (15 minutes of warm-up with slow walk, mobility and stretching exercise, followed by 30 minutes of a propioceptive exercises program, and finishing with 10 minutes of cool down through stretching and relaxation exercises)
  Arms: Experimental
Other: No propioceptive program — The control group continued to perform their daily activities without changing any habit. Geriatric revitalization program without proprioceptive exercises.
  Arms: Cotrol

SUMMARY:
Knowing the effects of proprioceptive exercise program in improving balance, gait and risk of falls in institutionalized elderly.

DETAILED DESCRIPTION:
The aim of this study will be to determine the effects of proprioceptive exercise program in improving balance and gait as well as reducing the risk of falls in institutionalized elderly in a healthcare center. To evaluate this effect, a total of 45 subjects will participate in a longitudinal and controlled trial. Inclusion criteria will be over 65 years olds, be institutionalized in the center and have ability to read and write.

Thereafter, participants will be separated into two different groups (experimental and control). Randomization was performed using sealed envelopes with different numbers of intervention inside. Both groups will be evaluated both at the start of the first session and in the last working session.

The control group performed a geriatric revitalization program as the experimental group. Besides this one, experimental group performed a program of proprioceptive exercises. The intervention rate will 2 weekly sessions for 12 weeks for both groups (24 sessions), lasting 55 minutes. The variables analyzed were: the questionnaire risk of falls in hospital (MORSE), Tinetti scale, the test Timed Up and Go (TUG), the time of one leg and the Cooper test running 12 minutes.

The data analysis will perform using the Statistical Package for the Social Sciences (SPSS statistical software), version 19.0 for Windows, Chicago.

To determine the normal distribution of the data the Shapiro-Wilks test and comparison by ANOVA was performed. The values obtained in the pretest and posttest assessment for each variable will be compared by Student t test for related samples or by the Wilcoxon rank test.

ELIGIBILITY:
Inclusion Criteria:

* Being institutionalized,
* own ability to read and write,
* and access the study voluntarily.

Exclusion Criteria:

* Significant degree of cognitive impairment;
* intolerance moderate physical activity, caused by cardiovascular or respiratory disease,
* as well as those who did not complete 90% of the sessions.

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Time Up and Go (TUG) test | Participants will be followed an expected average of 5 weeks.
  Evaluates mobility testing both static balance and the dynamic by measuring the time taken to perform a task.

SECONDARY OUTCOMES:
Tinnetti scale | Participants will be followed an expected average of 5 weeks.
  It consists of two subscales, gait and balance, where less than 19 points overall results indicate a high risk of falling
Questionnaire risk of falls in hospital (Morse) | Participants will be followed an expected average of 5 weeks.
  This questionnaire has 6 items with a total range of 0-125.
Cooper test | Participants will be followed an expected average of 5 weeks.
  Walking for 12 minutes around cones along the floor.
Support time monopodal | Participants will be followed an expected average of 5 weeks.
  Postural control is valued.

CONTACTS AND LOCATIONS:
Overall Officials: María Ángeles Cardero-Durán, PhD, Principal Investigator — University of Extremadura
Locations (1):
- Socio- Health Center Puente Real ( Health Care for Older © ) of Badajoz, Badajoz, Extremadura, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mather AS, Rodriguez C, Guthrie MF, McHarg AM, Reid IC, McMurdo ME. Effects of exercise on depressive symptoms in older adults with poorly responsive depressive disorder: randomised controlled trial. Br J Psychiatry. 2002 May;180:411-5. doi: 10.1192/bjp.180.5.411. PMID 11983637
- [Background] Geiger RA, Allen JB, O'Keefe J, Hicks RR. Balance and mobility following stroke: effects of physical therapy interventions with and without biofeedback/forceplate training. Phys Ther. 2001 Apr;81(4):995-1005. PMID 11276182
- [Background] Iwamoto J, Suzuki H, Tanaka K, Kumakubo T, Hirabayashi H, Miyazaki Y, Sato Y, Takeda T, Matsumoto H. Preventative effect of exercise against falls in the elderly: a randomized controlled trial. Osteoporos Int. 2009 Jul;20(7):1233-40. doi: 10.1007/s00198-008-0794-9. Epub 2008 Nov 15. PMID 19011727
- [Background] Stathokostas L, Little RM, Vandervoort AA, Paterson DH. Flexibility training and functional ability in older adults: a systematic review. J Aging Res. 2012;2012:306818. doi: 10.1155/2012/306818. Epub 2012 Nov 8. PMID 23209904
- [Result] Hewitt J, Refshauge KM, Goodall S, Henwood T, Clemson L. Does progressive resistance and balance exercise reduce falls in residential aged care? Randomized controlled trial protocol for the SUNBEAM program. Clin Interv Aging. 2014 Feb 21;9:369-76. doi: 10.2147/CIA.S53931. eCollection 2014. PMID 24591821
- [Result] Jorstad EC, Hauer K, Becker C, Lamb SE; ProFaNE Group. Measuring the psychological outcomes of falling: a systematic review. J Am Geriatr Soc. 2005 Mar;53(3):501-10. doi: 10.1111/j.1532-5415.2005.53172.x. PMID 15743297
- [Result] Howe TE, Rochester L, Neil F, Skelton DA, Ballinger C. Exercise for improving balance in older people. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD004963. doi: 10.1002/14651858.CD004963.pub3. PMID 22071817
- [Result] Sturnieks DL, Finch CF, Close JC, Tiedemann A, Lord SR, Pascoe DA. Exercise for falls prevention in older people: assessing the knowledge of exercise science students. J Sci Med Sport. 2010 Jan;13(1):59-64. doi: 10.1016/j.jsams.2008.11.005. Epub 2009 Feb 20. PMID 19230765
- [Result] Orr R, Raymond J, Fiatarone Singh M. Efficacy of progressive resistance training on balance performance in older adults : a systematic review of randomized controlled trials. Sports Med. 2008;38(4):317-43. doi: 10.2165/00007256-200838040-00004. PMID 18348591
- [Result] Cameron ID, Gillespie LD, Robertson MC, Murray GR, Hill KD, Cumming RG, Kerse N. Interventions for preventing falls in older people in care facilities and hospitals. Cochrane Database Syst Rev. 2012 Dec 12;12:CD005465. doi: 10.1002/14651858.CD005465.pub3. PMID 23235623
- [Result] Barnett A, Smith B, Lord SR, Williams M, Baumand A. Community-based group exercise improves balance and reduces falls in at-risk older people: a randomised controlled trial. Age Ageing. 2003 Jul;32(4):407-14. doi: 10.1093/ageing/32.4.407. PMID 12851185
- [Result] O'Connell B, Myers H. The sensitivity and specificity of the Morse Fall Scale in an acute care setting. J Clin Nurs. 2002 Jan;11(1):134-6. doi: 10.1046/j.1365-2702.2002.00578.x. No abstract available. PMID 11845750
- [Result] Tinetti ME, Williams TF, Mayewski R. Fall risk index for elderly patients based on number of chronic disabilities. Am J Med. 1986 Mar;80(3):429-34. doi: 10.1016/0002-9343(86)90717-5. PMID 3953620
- [Result] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Result] Vellas BJ, Wayne SJ, Romero L, Baumgartner RN, Rubenstein LZ, Garry PJ. One-leg balance is an important predictor of injurious falls in older persons. J Am Geriatr Soc. 1997 Jun;45(6):735-8. doi: 10.1111/j.1532-5415.1997.tb01479.x. PMID 9180669
- [Result] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Result] Banez C, Tully S, Amaral L, Kwan D, Kung A, Mak K, Moghabghab R, Alibhai SM. Development, implementation, and evaluation of an Interprofessional Falls Prevention Program for older adults. J Am Geriatr Soc. 2008 Aug;56(8):1549-55. doi: 10.1111/j.1532-5415.2008.01790.x. Epub 2008 Jun 28. PMID 18557964
- [Result] Espejo Antunez L, Cardero Duran MA, Caro Puertolas B, Tellez de Peralta G. [Effects of exercise on the function and quality of life in the institutionalised elderly diagnosed with gonarthrosis]. Rev Esp Geriatr Gerontol. 2012 Nov-Dec;47(6):262-5. doi: 10.1016/j.regg.2011.06.011. Epub 2012 May 14. Spanish. PMID 22592162
- [Derived] Espejo-Antunez L, Perez-Marmol JM, Cardero-Duran MLA, Toledo-Marhuenda JV, Albornoz-Cabello M. The Effect of Proprioceptive Exercises on Balance and Physical Function in Institutionalized Older Adults: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Oct;101(10):1780-1788. doi: 10.1016/j.apmr.2020.06.010. Epub 2020 Jul 12. PMID 32663479